CLINICAL TRIAL: NCT01399242
Title: Efficacy and Safety of Certican® in Combination With Myfortic® in Adult Renal Allograft Recipients Following Calcineurin Inhibitor Withdrawal at Week 16 Compared to Patients Who Are Maintained on Tacrolimus and Myfortic®
Brief Title: Efficacy of Certican® in Combination With Myfortic® in Renal
Acronym: HUSJ1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitário São José (Other)
Responsible Party: Euler Pace Lasmar, Hospital Universitário Sao Jose
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EL-1254
Record Dates: First submitted 2011-06-20; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-03

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Disorder Related to Renal Transplantation
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Certican, prednisona, EC-MPS (Active Comparator): Twenty patients will be selected at 16 weeks of renal transplantation to convert a immunosuppression to certican,prednisone and myfortic. The allocation will be done randomly to provide similar epidemiological characteristics with respect to gender, age, renal function and co morbidities in the two groups. The informed consent will obtained after an interview involving the researcher and patient when the protocol will be explained.A protocol renal biopsy will be performed at the end of the study, 12 months after transplantation
  Interventions: Drug: Certican
- Tacrolimus,Prednisona, EC-MPS (No Intervention): Twenty patients will be selected at 16 weeks of renal transplant to continue use EC-MPS,Tacrolimus and Prednisone. The allocation will be done randomly to provide similar epidemiological characteristics with respect to gender, age, renal function and co morbidities in the two groups. The informed consent will obtained after an interview involving the researcher and patient when the protocol will be explained.A protocol renal biopsy will be performed at the end of the study, 12 months after transplantation

INTERVENTIONS:
Drug: Certican — Patients' therapy will be replaced from tacrolimus-based to everolimus-based immunosuppression. Everolimus will be introduced on day 1 at dose of 2 mg/day (1mg bid), and then everolimus trough levels will be obtained from day 3 onwards until C0 reaches the target for three consecutive days. Through levels will be adjusted to achieve 6-10ng/ml. Thereafter, if the target level was reached, the measurement will be performed weekly for 4 weeks and every 2 weeks until 8 weeks after conversion.In parallel, the tacrolimus dose will be reduced by 50% on day 1 and another 25% on day 7. The Tacrolimus will be withdrawn on day 14 if the target levels of everolimus are obtained.EC-MPS will be unchanged until day 14 after conversion.
  Other Names: Myfortic, Prograf, Certican.
  Arms: Certican, prednisona, EC-MPS

SUMMARY:
The primary objective is to demonstrate the superiority of everolimus plus Myfortic® plus corticosteroids following CNI withdrawal at week 16 compared to tacrolimus plus Myfortic® plus corticosteroids as measured by the change in calculated Glomerular Filtration Rate (cGFR) from baseline to month 12.

The key secondary objective is to demonstrate non-inferiority of biopsy-proved acute rejection (BPAR), graft loss, death or loss to follow-up (composite endpoint) at month 12 in patients switched to everolimus plus Myfortic® plus corticosteroids following CNI withdrawal at Week 16 compared to patients maintained on tacrolimus plus Myfortic® plus corticosteroids.

Patients will be submitted to monthly GFR determination but, for group comparison, only the GFR measured at month 12 and month 24 of renal transplantation will be used.

DETAILED DESCRIPTION:
1.Forty patients will be selected at 16 weeks of renal transplantation with 20 patients allocated in each study arm. The allocation will be done randomly to provide similar epidemiological characteristics with respect to gender, age, renal function and co morbidities in the two groups. The informed consent will obtained after an interview involving the researcher and patient when the protocol will be explained.

1.1 Study protocol

Patients of renal transplant unit at the Sao Jose University Hospital who sign the inform consent and fulfill the inclusion/exclusion criteria will be enrolled in this study.

The main population will be low-risk kidney transplant recipients defined as follow: primary transplant, patients older than 18 years old and recipients of first kidney transplantation with living donor with PRA <10%, using tacrolimus, EC-MPS, and steroids as primary immunosuppression, without delayed graft function and with stable renal function 3 months after transplantation.

Patients who fulfill the inclusion criteria and agree to participate in this study will have the CNI withdrawn and the immunosuppressive regimen will be based on everolimus.

The switch will be done as follows: patients' therapy will be replaced from CNI-based to everolimus-based immunosuppression. Everolimus will be introduced on day 1 at dose of 2 mg/day (1mg bid), and then everolimus trough levels will be obtained from day 3 onwards until C0 reaches the target for three consecutive days. Through levels will be adjusted to achieve 6-10ng/ml. Thereafter, if the target level was reached, the measurement will be performed weekly for 4 weeks and every 2 weeks until 8 weeks after conversion.

In parallel, the CNI dose will be reduced by 50% on day 1 and another 25% on day 7. The CNI will be withdrawn on day 14 if the target levels of everolimus are obtained. EC-MPS will be unchanged until day 14 after conversion, thereafter it will be decreased if necessary from 1440mg to 1080mg/day. The dose of EC-MPS will not be below 1080 mg/day.

Corticosteroids would be unchanged. A protocol renal biopsy will be performed at the end of the study, 12 months after transplantation. A per-operatory biopsy at baseline will not be performed, since this is not a routine practice of the transplant center and because the patients have a low immunological risk.

1.3- Inclusion criteria

1.3.1- Men and women between 18-70 years old 1.3.2- Receptors of a first living-donor kidney allograft 1.3.3- Patients must have been on a tacrolimus+myfortic regimen for at least 2 weeks prior to randomization

1.4- Exclusion criteria

1.4.1- Patients with evidence of any acute rejection following transplantation at the time of randomization 1.4.2- GFR ≤ 35 ml/min 1.4.3- Proteinuria > 800 mg/day 1.4.4- Recipients of multiple organ transplants 1.4.5- Chronic hepatic failure 1.4.6- Asymptomatic bacteriuria 1.4.7- Creatinine ≥ 2mg/dL on CNI withdrawn time 1.4.8- Proteinuria ≥ 1g/24h on CNI withdrawn time 1.4.9- Presence of uncontrolled hypercholesterolemia (≥ 350 mg/dL, ≥ 9.1 mmol/L) 1.4.10- Hypertriglyceridemia (≥ 500 mg/dL, ≥ 5.6 mmol/L)

1.5- Statistical analysis

This is an investigational and interventional study, with two-arms, to evaluate the renal function and composite efficacy end-point after conversion of immunosuppressive regime from tacrolimus to everolimus. As this is a pilot study, the sample size was estimated with 20 patients in each arm (total = 40 patients) according to the number of kidney transplants usually performed at the hospital.

For GRF evaluation ANOVA will be used. A difference of 5-10ml/min at GRF is expected comparing study and control group.

The incidence of acute rejection will be analyzed by chi-square.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18-70 years old
* Receptors of a first living-donor kidney allograft
* Patients must have been on a tacrolimus+myfortic regimen for at least 2 weeks prior to randomization

Exclusion Criteria:

* Patients with evidence of any acute rejection following transplantation at the time of randomization
* GFR ≤ 35 ml/min
* Proteinuria > 800 mg/day
* Recipients of multiple organ transplants
* Chronic hepatic failure
* Asymptomatic bacteriuria
* Creatinine ≥ 2mg/dL on CNI withdrawn time
* Proteinuria ≥ 1g/24h on CNI withdrawn time
* Presence of uncontrolled hypercholesterolemia (≥ 350 mg/dL, ≥ 9.1 mmol/L)
* Hypertriglyceridemia (≥ 500 mg/dL, ≥ 5.6 mmol/L)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | 96 weeks
  The primary objective is to demonstrate the superiority of everolimus plus Myfortic® plus corticosteroids following CNI withdrawal at week 16 compared to tacrolimus plus Myfortic® plus corticosteroids as measured by the change in calculated Glomerular Filtration Rate (cGFR) from baseline to month 12.

SECONDARY OUTCOMES:
Non-inferiority of biopsy-proved acute rejection (BPAR), graft loss, death | 1 year after enrollment
  The key secondary objective is to demonstrate non-inferiority of biopsy-proved acute rejection (BPAR), graft loss, death or loss to follow-up (composite endpoint) at month 12 in patients switched to everolimus plus Myfortic® plus corticosteroids following CNI withdrawal at Week 16 compared to patients maintained on tacrolimus plus Myfortic® plus corticosteroids.

CONTACTS AND LOCATIONS:
Overall Officials: Euler P lasmar, Study Director — Hospital Universitário Sao José
Locations (1):
- Hospital Universitário São José, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Pilmore HL, Dittmer ID. Calcineurin inhibitor nephrotoxicity: reduction in dose results in marked improvement in renal function in patients with coexisting chronic allograft nephropathy. Clin Transplant. 2002 Jun;16(3):191-5. doi: 10.1034/j.1399-0012.2002.01119.x. PMID 12010142
- [Background] Mendez R, Gonwa T, Yang HC, Weinstein S, Jensik S, Steinberg S; Prograf Study Group. A prospective, randomized trial of tacrolimus in combination with sirolimus or mycophenolate mofetil in kidney transplantation: results at 1 year. Transplantation. 2005 Aug 15;80(3):303-9. doi: 10.1097/01.tp.0000167757.63922.42. PMID 16082323
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Lorber MI, Mulgaonkar S, Butt KM, Elkhammas E, Mendez R, Rajagopalan PR, Kahan B, Sollinger H, Li Y, Cretin N, Tedesco H; B251 Study Group. Everolimus versus mycophenolate mofetil in the prevention of rejection in de novo renal transplant recipients: a 3-year randomized, multicenter, phase III study. Transplantation. 2005 Jul 27;80(2):244-52. doi: 10.1097/01.tp.0000164352.65613.24. PMID 16041270
- [Background] Johnson RW. The clinical impact of nephrotoxicity in renal transplantation. Transplantation. 2000 Jun 27;69(12 Suppl):SS14-7. doi: 10.1097/00007890-200006271-00004. No abstract available. PMID 10910258
- [Background] Gallon L, Perico N, Dimitrov BD, Winoto J, Remuzzi G, Leventhal J, Gaspari F, Kaufman D. Long-term renal allograft function on a tacrolimus-based, pred-free maintenance immunosuppression comparing sirolimus vs. MMF. Am J Transplant. 2006 Jul;6(7):1617-23. doi: 10.1111/j.1600-6143.2006.01340.x. PMID 16827862
- [Background] Tedesco-Silva H Jr, Vitko S, Pascual J, Eris J, Magee JC, Whelchel J, Civati G, Campbell S, Alves-Filho G, Bourbigot B, Garcia VD, Leone J, Esmeraldo R, Rigotti P, Cambi V, Haas T; 2306 and 2307 study groups. 12-month safety and efficacy of everolimus with reduced exposure cyclosporine in de novo renal transplant recipients. Transpl Int. 2007 Jan;20(1):27-36. doi: 10.1111/j.1432-2277.2006.00414.x. PMID 17181650
- [Background] Ciancio G, Burke GW, Gaynor JJ, Mattiazzi A, Roth D, Kupin W, Nicolas M, Ruiz P, Rosen A, Miller J. A randomized long-term trial of tacrolimus and sirolimus versus tacrolimus and mycophenolate mofetil versus cyclosporine (NEORAL) and sirolimus in renal transplantation. I. Drug interactions and rejection at one year. Transplantation. 2004 Jan 27;77(2):244-51. doi: 10.1097/01.TP.0000101290.20629.DC. PMID 14742989
- [Background] Ciancio G, Burke GW, Gaynor JJ, Ruiz P, Roth D, Kupin W, Rosen A, Miller J. A randomized long-term trial of tacrolimus/sirolimus versus tacrolimums/mycophenolate versus cyclosporine/sirolimus in renal transplantation: three-year analysis. Transplantation. 2006 Mar 27;81(6):845-52. doi: 10.1097/01.tp.0000203894.53714.27. PMID 16570006
- [Background] Ciancio G, Burke GW, Gaynor JJ, Mattiazzi A, Roth D, Kupin W, Nicolas M, Ruiz P, Rosen A, Miller J. A randomized long-term trial of tacrolimus/sirolimus versus tacrolimus/mycophenolate mofetil versus cyclosporine (NEORAL)/sirolimus in renal transplantation. II. Survival, function, and protocol compliance at 1 year. Transplantation. 2004 Jan 27;77(2):252-8. doi: 10.1097/01.TP.0000101495.22734.07. PMID 14742990